CLINICAL TRIAL: NCT00003678
Title: A Large, Uniquely Simple, Randomised Study to Assess Much More Reliably the Balance of Benefits and Risks of Prolonging Adjuvant Tamoxifen Treatment in Early Breast Cancer
Brief Title: Tamoxifen in Treating Women With Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Birmingham (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066779; CRC-TU-ATTOM; EU-98042; ISRCTN17222211
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: tamoxifen citrate
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking the uptake of estrogen by the tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of at least 2 years of tamoxifen with that of 5 additional years of tamoxifen in treating women who have breast cancer that has been surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free and overall survival of women with early breast cancer who are randomized to discontinue adjuvant tamoxifen vs those randomized to continue for at least 5 additional years.

OUTLINE: This is a randomized study. Patients are stratified for analysis according to duration of tamoxifen given before randomization (2-3 years vs 4-5 years vs 6-7 years vs 8-9 years vs 10 years and over), age (less than 49 vs over 50), and important prognostic factors, including tumor type and grade and nodal and estrogen receptor status. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients discontinue tamoxifen after at least 2 years of prior treatment.
* Arm II: Patients continue treatment with tamoxifen for at least 5 additional years in the absence of unacceptable toxicity or disease progression.

Patients are followed annually.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 8,000-20,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast carcinoma that has been completely excised

  * Clinically relapse free
* Must have completed at least two years of adjuvant therapy with tamoxifen for early breast cancer AND have no clear indication for or against receiving further tamoxifen
* No significant endometrial hyperplasia
* No patients with negligibly low risk of breast cancer death
* Hormone receptor status:

  * Any status allowed

PATIENT CHARACTERISTICS:

Age:

* Not specified

Sex:

* Female

Menopausal status:

* Any status allowed

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other life threatening disease
* No retinopathy
* No psychiatric disorder or other condition that would preclude study compliance
* No serious toxicity (e.g., depression) thought to be due to tamoxifen
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* Any primary treatment allowed

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 1991-05

PRIMARY OUTCOMES:
All-cause mortality

SECONDARY OUTCOMES:
Disease recurrence
Death due to breast cancer, other primary tumors, or cardiovascular causes

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rea, MD, Study Chair — University Hospital Birmingham
Locations (1):
- Cancer Research UK Clinical Trials Unit - Birmingham, Birmingham, England, United Kingdom

REFERENCES:
- [Background] Gray R, Davies C, Perry P. Tamoxifen for early breast cancer: better late than never. Ann Oncol. 2000 May;11(5):505-7. doi: 10.1023/a:1008323116265. No abstract available. PMID 10907940
- [Background] Rea D, Poole C, Gray R. Adjuvant tamoxifen: how long before we know how long? BMJ. 1998 May 16;316(7143):1518-9. doi: 10.1136/bmj.316.7143.1518. No abstract available. PMID 9582148
- [Background] Earl H, Gray R, Kerr D, Lee M. The optimal duration of adjuvant tamoxifen treatment for breast cancer remains uncertain: randomize into aTTom. Clin Oncol (R Coll Radiol). 1997;9(3):141-3. doi: 10.1016/s0936-6555(97)80067-2. No abstract available. PMID 9269542
- [Background] Earl H, Baker P, Kerr D, Lee M, Gray R, Baum M. Adjuvant treatment with tamoxifen. Recruitment into studies assessing optimum duration of treatment must continue. BMJ. 1996 Apr 20;312(7037):1036-7. doi: 10.1136/bmj.312.7037.1036b. No abstract available. PMID 8616358
- [Background] Gray R. Tamoxifen: how boldly to go where no women have gone before. J Natl Cancer Inst. 1993 Sep 1;85(17):1358-60. doi: 10.1093/jnci/85.17.1358. No abstract available. PMID 8350355
- [Derived] Poterala JE, Wisinski KB. Abbreviated endocrine therapy duration for low estrogen receptor-positive breast cancer: The counter to extended endocrine therapy. Cancer. 2022 May 1;128(9):1724-1726. doi: 10.1002/cncr.34158. Epub 2022 Feb 25. No abstract available. PMID 35213039
- [Derived] Bartlett JMS, Sgroi DC, Treuner K, Zhang Y, Ahmed I, Piper T, Salunga R, Brachtel EF, Pirrie SJ, Schnabel CA, Rea DW. Breast Cancer Index and prediction of benefit from extended endocrine therapy in breast cancer patients treated in the Adjuvant Tamoxifen-To Offer More? (aTTom) trial. Ann Oncol. 2019 Nov 1;30(11):1776-1783. doi: 10.1093/annonc/mdz289. PMID 31504126